CLINICAL TRIAL: NCT00554840
Title: Comparison of Varenicline and Placebo for Smoking Cessation in Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, MPRC, Physician, Maryland Psychiatric Research Center, Outpatient Research Program, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-00042225
Record Dates: First submitted 2007-11-06; First posted 2007-11-07 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Cigarette Smoking; Schizophrenia
MeSH Terms: conditions — Cigarette Smoking; Schizophrenia | interventions — Varenicline; Drug Evaluation; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- varenicline (Active Comparator)
  Interventions: Drug: varenicline
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: varenicline — Subjects will be randomized to receive either active drug or matching placebo capsules using the following titration schedule: 0.5mg for three days, 0.5mg twice daily for the next four days, then 1mg twice daily for the rest of the treatment phase. Subjects will be evaluated weekly for abstinence through self report, end expired CO and urine dipstick for cotinine.
  Other Names: chantix, study drug
  Arms: varenicline
Drug: placebo — At the end of Pre-med week 1, subjects will receive study medication with the target quit date being the following week. Subjects will be randomized to receive either active drug or matching placebo capsules using the following titration schedule: 0.5mg for three days, 0.5mg twice daily for the next four days, then 1mg twice daily for the rest of the treatment phase. Subjects will be evaluated weekly for abstinence through self report, end expired CO and urine dipstick for cotinine.
  Other Names: sugar pill
  Arms: placebo

SUMMARY:
The purpose of this proposed pilot study is to examine the use of varenicline in people with schizophrenia to specifically assess tolerability and efficacy for smoking cessation. Specifically, The primary objective of this pilot study is to determine if taking of varenicline along with an individual smoking cessation supportive program is a safe and effective treatment of nicotine addiction in schizophrenic patients. We hypothesize that the varenicline treated patients will achieve higher rates of smoking cessation than those who receive placebo and individual support.

DETAILED DESCRIPTION:
The primary objective of the data analysis will be to measure the rate of smoking cessation in the two treatment groups. Smoking cessation will be measured weekly through a composite measure of self-reported abstinence, end expired carbon monoxide (CO) of less than C10 ppm and urine cotinine dipstick measure of < 30 ng/ml. The primary endpoint will be point prevalence at 12 weeks. The four week continuous abstinence rate for the last four weeks of the treatment phase will also be evaluated. The point prevalence abstinence rates will also be obtained. The secondary objective is to determine whether smoking cessation is associated with a worsening of cognition and psychiatric symptomology. We hypothesize that subjects who achieve abstinence in the varenicline group will not show worsening on neurocognitive and symptom measures compared to abstinence subjects in the placebo group. Lastly, we will attempt to identify any clinical or topographic markers which predict cessation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-64
* Regular ten cigarette per day smoker for one year
* Nicotine Dependency Score greater than or equal to four
* DSM-IV Diagnosis of Schizophrenia or Schizoaffective disorder
* Psychiatric medication regimen unchanged for at least 90 days
* Psychiatric medication dosage unchanged for at least 30 days

Exclusion Criteria:

* Psychiatric hospitalization in last 6 months
* Meets criteria for current Major Depressive Disorder or has a score of greater than 10 on the Calgary Depression Scale (see withdrawal criteria)
* Suicide or homicide ideation with a plan in the last six months
* Life time history of suicide attempt
* Has had a diagnosis of Schizophrenia or Schizoaffective disorder for less than three years
* Current treatment with Bupropion SR
* DSM-IV diagnosis of alcohol or substance dependence within last 6 months*
* DSM-IV diagnosis of alcohol or substance abuse within three months *
* Pregnancy or lactation in females (+HCG)
* Use of tobacco product other than cigarettes
* Use of nicotine replacements
* Unstable or serious medical condition in last 6 months
* Regular use of cimetidine (OTC or Rx) *Substance abuse/dependency exclusions do not apply to abuse of or dependence on nicotine.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2007-11; Primary Completion 2010-12 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Weiner, M.D., Principal Investigator — Maryland Psychiatric Research Center

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Stable outpatients who received their regular treatment at the Outpatient Research Program of the MPRC were invited to participate.
Pre-assignment Details: After the enrollment of 16 participants, a total of 7 participants were withdrawn from the study prior to assignment to a treatment group (n=9). Two subjects met exclusion criteria before any study procedures were started, and 5 subjects were withdrawn during either the "evaluation" or "pre-med" phases of the study.
Period: Overall Study
Arm/Group | Varenicline | Placebo
Started | 4 | 5
Completed | 4 | 4
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: One participant was withdrawn by the P.I. after assignment to the placebo group, but prior to receiving treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (9.0) | 44.3 (5.1) | 45.97 (6.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 3 | 6
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change of ExpiredCO Level From Baseline
Description: End expired carbon monoxide (CO) level change from baseline to determine participants' level of smoking reduction by treatment assignment. Larger negative values represent a greater level of smoking reduction.
Time Frame: Weekly for 12 weeks
Population: Some ExpiredCO data is missing due to rater error or participant absence from that study visit.
Measure: Mean (Standard Deviation); unit: ppm
Groups:
- Varenicline: Subjects randomized to active treatment (varenicline) will use the following titration schedule: 0.5mg for three days, 0.5mg twice daily for the next four days, then 1mg twice daily for the rest of the treatment phase.
- Placebo: Subjects randomized to matching placebo capsules will use the following titration schedule: 0.5mg for three days, 0.5mg twice daily for the next four days, then 1mg twice daily for the rest of the treatment phase.
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 4 | 4
ppm
  Treatment Week 1 | -2.88 (8.35) | 9.5 (6.54)
  Treatment Week 2 | -17.38 (22.21) | -11.5 (6.94)
  Treatment Week 3 | -17.13 (23.59) | -5.75 (2.40)
  Treatment Week 4 | -18.63 (20.77) | 2.5 (4.10)
  Treatment Week 5 | -20.63 (20.27) | -4.5 (4.02)
  Treatment Week 6: number analyzed (Participants) | 4 | 3
  Treatment Week 6 | -20.38 (20.55) | -3.83 (7.25)
  Treatment Week 7: number analyzed (Participants) | 4 | 3
  Treatment Week 7 | -20.13 (20.46) | -2.83 (7.11)
  Treatment Week 8: number analyzed (Participants) | 4 | 3
  Treatment Week 8 | -20.88 (19.28) | -4.83 (8.40)
  Treatment Week 9: number analyzed (Participants) | 4 | 3
  Treatment Week 9 | -20.88 (19.98) | -0.17 (12.55)
  Treatment Week 10: number analyzed (Participants) | 4 | 3
  Treatment Week 10 | -21.13 (19.38) | -2.83 (9.78)
  Treatment Week 11: number analyzed (Participants) | 4 | 3
  Treatment Week 11 | -19.63 (20.72) | 8.17 (17.19)
  Treatment Week 12 | -19.875 (18.98) | -0.75 (6.64)

2. Primary Outcome: Level of Nicotine Dependence by Treatment Assignment
Description: Nicotine dependence was measured using the total score from the Fagerstrom Test for Nicotine Dependence (FTND) assessment. The total score is computed by adding the scores from the five subscales. Total scores range from 1-10, with lower scores representing a smaller degree of nicotine dependence.
Time Frame: Weekly for 12 weeks
Population: Some FTND data is missing due to rater error or participant absence from that study visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 4 | 4
units on a scale
  Treatment Week 0 | 5.88 (1.31) | 5.75 (2.10)
  Treatment Week 1 | 4.5 (1.30) | 5.25 (2.06)
  Treatment Week 2: number analyzed (Participants) | 3 | 4
  Treatment Week 2 | 4.33 (0.58) | 4.75 (2.06)
  Treatment Week 3: number analyzed (Participants) | 3 | 4
  Treatment Week 3 | 3 (3) | 4.5 (1.91)
  Treatment Week 4: number analyzed (Participants) | 3 | 4
  Treatment Week 4 | 3 (3) | 5 (1.83)
  Treatment Week 5 | 2.75 (2.22) | 5.25 (1.71)
  Treatment Week 6: number analyzed (Participants) | 4 | 3
  Treatment Week 6 | 4.25 (1.71) | 4.33 (1.53)
  Treatment Week 7: number analyzed (Participants) | 4 | 3
  Treatment Week 7 | 4.5 (1.73) | 4.67 (1.53)
  Treatment Week 8: number analyzed (Participants) | 4 | 3
  Treatment Week 8 | 4.75 (1.89) | 4 (1.73)
  Treatment Week 9: number analyzed (Participants) | 4 | 3
  Treatment Week 9 | 5 (2.16) | 3.67 (2.08)
  Treatment Week 10: number analyzed (Participants) | 4 | 3
  Treatment Week 10 | 5 (2) | 3.67 (2.08)
  Treatment Week 11: number analyzed (Participants) | 3 | 3
  Treatment Week 11 | 6 (1) | 4.33 (1.53)
  Treatment Week 12 | 3.5 (3.11) | 4.25 (1.5)

3. Secondary Outcome: Brief Psychiatric Rating Scale (BPRS) - Total Score
Description: The total BPRS score is calculated by adding the scores for subscales #1-#18. Each scale ranges from "1=Not Present" to "7=Very Severe". Total scores range from a minimum score of 18 to a maximum score of 126. A higher total score indicates a more severe psychiatric symptom rating.
Time Frame: Baseline (week 0) then again during the Treatment Phase at weeks 1, 2, 4, 8, and 12.
Population: Some BPRS total score data is missing due to rater error or participant absence from that study visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 4 | 4
units on a scale
  Baseline | 35.75 (6.34) | 30.25 (4.11)
  Treatment Week 1 | 33.75 (5.56) | 32.75 (6.6)
  Treatment Week 2 | 35.5 (7) | 30.25 (4.35)
  Treatment Week 4 | 31.75 (3.4) | 30.25 (6.75)
  Treatment Week 8: number analyzed (Participants) | 4 | 3
  Treatment Week 8 | 36.25 (4.27) | 28 (2.65)
  Treatment Week 12 | 34.75 (3.30) | 32 (3.92)

4. Secondary Outcome: Brief Psychiatric Rating Scale (BPRS) - Psychosis Score
Description: The psychosis score is calculated by adding the scores for scales #4 Conceptual Disorganization, #11 Suspiciousness, #12 Hallucinatory Behavior, and #15 Unusual Thought Content. Each scale ranges from "1=Not Present" to "7=Very Severe". The minimum psychosis score is 4 and the maximum psychosis score is 28. A higher score indicates a more severe psychosis rating.
Time Frame: Baseline (week 0) then again during the Treatment Phase at weeks 1, 2, 4, 8, and 12.
Population: Some BPRS total score data is missing due to rater error or participant absence from that study visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 4 | 4
units on a scale
  Baseline | 11.25 (2.22) | 10 (5.94)
  Treatment Week 1 | 8.5 (3.12) | 11.5 (6.03)
  Treatment Week 2 | 9.25 (4.03) | 8.5 (4.51)
  Treatment Week 4 | 8.25 (4.03) | 8.5 (4.65)
  Treatment Week 8: number analyzed (Participants) | 4 | 3
  Treatment Week 8 | 10.75 (3.3) | 7.67 (1.53)
  Treatment Week 12 | 8.75 (2.22) | 10.5 (3.87)

5. Secondary Outcome: Brief Psychiatric Rating Scale (BPRS) - Anxiety/Depression Score
Description: The anxiety/depression score is calculated by adding the scores for scales #2 Anxiety and #9 Depressive Mood. Each scale ranges from "1=Not Present" to "7=Very Severe". The minimum anxiety/depression score is 2 and the maximum psychosis score is 14. A higher score indicates a more severe anxiety/depression rating.
Time Frame: Baseline (week 0) then again during the Treatment Phase at weeks 1, 2, 4, 8, and 12.
Population: Some BPRS anxiety/depression score data is missing due to rater error or participant absence from that study visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 4 | 4
units on a scale
  Baseline | 5.5 (1.3) | 6.75 (2.06)
  Treatment Week 1 | 3.25 (0.96) | 8 (3.27)
  Treatment Week 2 | 7.25 (1.71) | 7.25 (2.99)
  Treatment Week 4 | 6.25 (1.71) | 8 (4.32)
  Treatment Week 8: number analyzed (Participants) | 4 | 3
  Treatment Week 8 | 7.25 (0.5) | 3.37 (2.52)
  Treatment Week 12 | 7 (1.41) | 7.5 (2.65)

6. Secondary Outcome: Side Effects
Description: Side effects (33 items) were measured using a Side Effects Checklist (SEC). The percentage of participants endorsing each side effect were reported regardless of the severity or relation to study drug.
Time Frame: Weekly for 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 4 | 4
Participants
  Abdominal pain | 1 | 4
  Anorexia | 0 | 1
  Bruising | 0 | 0
  Constipation | 2 | 0
  Diarrhea | 1 | 0
  Dizziness | 1 | 2
  Dry mouth | 0 | 2
  Enuresis | 0 | 2
  Fever | 0 | 0
  Headache | 1 | 1
  Insomnia | 3 | 1
  Malaise | 2 | 1
  Mucosal ulceration | 0 | 0
  Nausea | 3 | 1
  Rash | 1 | 1
  Restlessness | 0 | 1
  Hypersalivation | 3 | 1
  Sedation | 2 | 2
  Stiffness | 0 | 1
  Sore throat | 1 | 1
  Tremor | 0 | 1
  Uticaria | 1 | 1
  Vomiting | 0 | 1
  Weight loss | 1 | 0
  Tinnitus | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each participant for their entire duration of the study (up to 20 weeks).
Groups:
- Varenicline: Subjects randomized to receive active drug (varenicline) will have the following titration schedule: 0.5mg for three days, 0.5mg twice daily for the next four days, then 1mg twice daily for the rest of the treatment phase.
- Placebo: Subjects randomized to matching placebo will have the following titration schedule: 0.5mg for three days, 0.5mg twice daily for the next four days, then 1mg twice daily for the rest of the treatment phase.
Arm/Group | Varenicline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/4
Other Adverse Events (participants affected / at risk) | 3/4 | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=4) | Placebo (N=4)
Hospitalization (Psychiatric disorders) | 0 (0) | 1 (1) — One subject was taken to the ER after exhibiting anxiety symptoms. This participant had a long history of going to the emergency room when he feels anxious due to worsening of anxiety, therefore, it is unlikely that the SAE was study drug related.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=4) | Placebo (N=4)
Dizziness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 0 (0)
Dry mouth (General disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Elevated liver enzymes (Hepatobiliary disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (3) | 0 (0)
Abdominal pain (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Larger studies are needed to confirm these encouraging results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes